CLINICAL TRIAL: NCT03790410
Title: The Effect of Inspiratory Muscle Training on Postural Control in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Levente Szilagyi, University Lecturer, Szeged University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COPD IMT PC
Record Dates: First submitted 2018-12-20; First posted 2018-12-31 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: COPD Postural Control IMT
Keywords: COPD Postural Control IMT

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group-Complex pulmonary rehab. (Active Comparator): Complex pulmonary rehabilitation:
  The complex pulmonary rehabilitation program containing breathing exercises, bicycle ergometer conditionings, relaxations, strength and endurance trainings.
  Interventions: Other: Complex pulmonary rehabilitation
- Inspiratory muscle training group (Active Comparator): Complex pulmonary rehabilitation:
  The complex pulmonary rehabilitation program containing breathing exercises, bicycle ergometer conditionings, relaxations, strength and endurance trainings.
  Inspiratory muscle training
  The training program contains strengthening exercises on the diaphragm muscle.
  Interventions: Other: Complex pulmonary rehabilitation; Other: Inspiratory muscle training

INTERVENTIONS:
Other: Complex pulmonary rehabilitation — Complex pulmonary rehabilitation program containing breathing exercises, bicycle ergometer conditionings, relaxations, strength and endurance trainings.
Other: Inspiratory muscle training — The training program contains strengthening exercises on the diaphragm muscle.
  Arms: Inspiratory muscle training group

SUMMARY:
Deficits in postural control are increasingly recognized among the important secondary impairments in patients with chronic obstructive pulmonary disease (COPD). There are conflicting results regarding the effect of inspiratory muscle training in improvement of inspiratory muscle strength, endurance, and dyspnea in stable COPD patients. The main inspiratory muscle, the diaphragm has also a stabilizing function of the trunk. The aim of this study to enhance postural control of COPD patients with improving the stability of the trunk by using inspiratory muscle training.

DETAILED DESCRIPTION:
The study is a randomized controlled trial in patients with stable COPD. The participants are divided into two groups. Patients in the inspiratory muscle training (IMT) group take part in a complex pulmonary rehabilitation program containing breathing exercises, bicycle ergometer conditionings, relaxations, strength and endurance trainings completed by inspiratory muscle training. The members of the IMT group use the POWERbreathe Medic device. The control group perform the complex pulmonary rehabilitation program without IMT. The program is divided into 3 weeks inpatient period and 3 weeks home period. Before, between and after the 3 weeks period all subjects are measured. 60 patients are planned to take part in the investigation. The inspiratory muscle strength is measured by POWERbreathe K1 device. Balance is assessed by functional balance tests: Timed Up and Go Test, Four Square Step Test, Modified Functional Reach Test, Modified Lateral Reach Test, Stand Up Test. Body Sway is measured by HR Mat VersaTek System. The diameter of the diaphragm muscle is assessed by B-mode ultrasound examination using Zonare Z. One Ultrasound System. Arterial stiffness parameters measured by Arteriograph.

ELIGIBILITY:
Inclusion Criteria:

* Stable COPD
* Do not take part in other treatment
* Be able to learn the usage of inspiratory muscle trainer

Exclusion Criteria:

* Acute exacerbation
* Balance problems with neurological cause
* The patient unable to cooperate
* Participation in pulmonary rehabilitation 3 months before the study
* IMT use in the 3 months before the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure | 6 weeks
  The inspiratory pressure generated against a completely occluded airway; used to evaluate inspiratory respiratory muscle strength and readiness for weaning from A maximum inspiratory pressure is measured in H2Ocm. MIP is measured with POWERbreathe K1
Timed Up and Go Test | 6 weeks
  Timed Up and Go: It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Four Square Step Test | 6 weeks
  Four Square Step Test:
  The subject is required to sequentially step over four canes set-up in a cross configuration on the ground. The aim is to step as fast as possible into each square with both feet.
Modified Functional Reach Test | 6 weeks
  Modified Functional Reach Test:
  The MFRT assesses a patient's stability by measuring the maximum distance an individual can reach forward while sitting in a fixed position.
Modified Lateral Reach Test | 6 weeks
  Modified Lateral Reach Test:
  The MLRT assesses a patient's stability by measuring the maximum distance an individual can reach side direction while sitting in a fixed position.
Stand Up Test | 6 weeks
  Stand Up Test:
  Individual stand up from tailor sit from the floor as fast as possible.

SECONDARY OUTCOMES:
Sway analysis: COF area (cm2) | 6 weeks
  Sway is the oscillating movement of the body, while posture is the relative alignment and orientation of the segments of the body. Sway analysis is a systematic assessment of the readiness and stability of the human body to achieve and maintain equilibrium. Area and direction of sway, elliptical pattern of sway, distance and direction traveled by Center of Force (CoF) is measured with HR Mat VersaTek System.
Sway analysis: COF distance (cm) | 6 weeks
  Sway is the oscillating movement of the body, while posture is the relative alignment and orientation of the segments of the body. Sway analysis is a systematic assessment of the readiness and stability of the human body to achieve and maintain equilibrium. Area and direction of sway, elliptical pattern of sway, distance and direction traveled by Center of Force (CoF) is measured with HR Mat VersaTek System.
Sway analysis: COF variability (cm) | 6 weeks
  Sway is the oscillating movement of the body, while posture is the relative alignment and orientation of the segments of the body. Sway analysis is a systematic assessment of the readiness and stability of the human body to achieve and maintain equilibrium. Area and direction of sway, elliptical pattern of sway, distance and direction traveled by Center of Force (CoF) is measured with HR Mat VersaTek System.
Sway analysis: COF A-P excursion (cm) | 6 weeks
  Sway is the oscillating movement of the body, while posture is the relative alignment and orientation of the segments of the body. Sway analysis is a systematic assessment of the readiness and stability of the human body to achieve and maintain equilibrium. Area and direction of sway, elliptical pattern of sway, distance and direction traveled by Center of Force (CoF) is measured with HR Mat VersaTek System.
Sway analysis: COF L-R excursion (cm) | 6 weeks
  Sway is the oscillating movement of the body, while posture is the relative alignment and orientation of the segments of the body. Sway analysis is a systematic assessment of the readiness and stability of the human body to achieve and maintain equilibrium. Area and direction of sway, elliptical pattern of sway, distance and direction traveled by Center of Force (CoF) is measured with HR Mat VersaTek System.
Thickness of the diaphragm muscle's belly | 6 weeks
  The diameter of the diaphragm muscle is assessed by B-mode ultrasound examination using Zonare Z. One Ultrasound System.
Vibration Sense Testing | 6 weeks
  Tuning fork is used to evaluate the deep sensation.
Pulse wave velocity | 6 weeks
  Pulse wave velocity is measured with Arteriograph.
Augmentation index | 6 weeks
  Augmentation index is measured with Arteriograph

CONTACTS AND LOCATIONS:
Locations (1):
- University of Szeged, Szeged, Csongrád megye, Hungary